CLINICAL TRIAL: NCT03737539
Title: Dynamic Monitoring of Circulating Tumor DNA Methylation to Predict Relapse in Colorectal Cancer After Radical Resection: A Prospective, Multicenter, Clinical Study (POSTCA)
Brief Title: Dynamic Monitoring of ctDNA Methylation to Predict Relapse in Colorectal Cancer After Radical Resection (POSTCA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Second Military Medical University (Other); Shanghai University of Traditional Chinese Medicine (Other); RenJi Hospital (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Professor, Fudan University
Other Study IDs: FDCRC42-CGX (POSTCA trial)
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Circulating Tumor DNA; Surveillance; Methylation
Keywords: Colorectal Cancer; Circulating tumor DNA; Surveillance; ctDNA Methylation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer: Patients diagnosed with resectable colorectal cancer
  Interventions: Diagnostic Test: Multigene methylation detection

INTERVENTIONS:
Diagnostic Test: Multigene methylation detection — Colorectal tumor-specific plasma ctDNA methylation markers detection

SUMMARY:
This is a prospective, multicenter, observational, single-blinded controlled study. Dynamic monitoring of patients with resectable colorectal cancer was performed using the previously established colorectal tumor-specific plasma ctDNA methylation markers (Multigene methylation detection). Dynamic monitoring of plasma ctDNA methylation before and after treatment and at regular follow-up in patients with colorectal cancer after radical resection of tumor, to explore the predictive effect of postoperative plasma ctDNA methylation on postoperative recurrence and whether dynamic monitoring of postoperative ctDNA methylation could be earlier than imaging examination to indicate tumor recurrence.

DETAILED DESCRIPTION:
At present, the main treatment of colorectal cancer (CRC) is surgical resection. CRC patients after radical surgery have good overall survival. However, there are still a large number of patients with postoperative recurrence. The postoperative recurrence rate of stage II CRC patients is 20-30%, and that of stage III CRC patients is 50-60%. Currently, there is no effective measures to predict whether patients suffer postoperative relapse. Patients can only periodically visit doctors in the hope of timely treatment in case of recurrence. Current clinical monitoring methods mainly include imaging detection and tumor markers detection. However, long-term monitoring may affect patients' quality of life and increase patients' economic burden. Therefore, biomarkers that can predict the prognosis of patients and screen out those who need intensive follow up are urgently warranted. At present, imaging is the mainly used approach to monitor tumor recurrence. Quantitative determination of ctDNA methylation in plasma may find tumor recurrence trend before imaging detection, indicating that quantitative determination of ctDNA methylation in plasma is a more sensitive monitoring approach than traditional imaging detection. Can plasma ctDNA methylation be a new recurrence monitoring technique and prognostic prediction method of CRC in clinical practice? In this study, we aimed to monitor the dynamic level of plasma ctDNA methylation after surgery in CRC patients, and to explore the advantages of plasma ctDNA methylation detection over traditional CRC in recurrence monitoring and prognosis prediction. This is a prospective, multicenter, observational, single-blinded controlled study. Dynamic monitoring of CRC patients was performed using the previously established colorectal tumor-specific plasma ctDNA methylation markers. Dynamic monitoring of plasma ctDNA methylation before and after treatment and at regular follow-up in patients with CRC after radical resection of tumor, to explore the predictive effect of postoperative plasma ctDNA methylation on postoperative recurrence and whether dynamic monitoring of postoperative ctDNA methylation could be earlier than imaging examination to indicate tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age on the day of signing informed consent.
* Patients must have histologically confirmed colorectal cancer.
* Patients need to receive surgical resection.
* Patients must have a performance status of ≤1 on the ECOG Performance Scale.
* Life expectancy of more than 5 years.
* Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

* Patients received adjuvant treatment prior to the surgical resection.
* Patients received blood transfusion two weeks before or during the surgical resection.
* Patients with unresected advanced colorectal adenoma.
* Patients who are positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C.
* Patients who are pregnant.
* Patients who are alcoholic or drug abusers.
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable colorectal cancer must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 2-year DFS
  The primary endpoint for this study is Disease Free Survival (DFS), which will be assessed using RECIST version 1.1.
ctDNA methylation markers versus CT/MRI | 2 years
  ctDNA methylation predictors of outcome will be compared to CT/MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China